CLINICAL TRIAL: NCT01519895
Title: Effectiveness of Telephone-based Intervention on Distress, Burden and Quality of Life of Chinese Caregivers of Colorectal Cancer Patients
Brief Title: Effectiveness of Telephone Intervention for Colorectal Cancer Caregivers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital Authority, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Shum Nga Fan, Department of Surgery, Colorectal Specialist Nurse, Principal Investigator, Hospital Authority, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HKCTR-1336
Record Dates: First submitted 2012-01-11; First posted 2012-01-27 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Psychological Stress
Keywords: quality of life; anxiety; stress; carers; colorectal or colon cancer
MeSH Terms: conditions — Stress, Psychological; Anxiety Disorders; Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Existing care (No Intervention): routine existing care
- Telephone intervention (Experimental): in addition to provide telephone intervention support
  Interventions: Behavioral: Telephone intervention

INTERVENTIONS:
Behavioral: Telephone intervention — counseling and education support
  Arms: Telephone intervention

SUMMARY:
The purpose of this study is to assess the effectiveness of the telephone intervention program for caregivers of colorectal cancer.

DETAILED DESCRIPTION:
telephone Intervention refer to provide counseling and education to caregivers of colorectal cancer by mode of telephone

ELIGIBILITY:
Inclusion Criteria:

* Family members with newly diagnosed colorectal cancer within the past 4 week and treated in Queen Mary Hospital
* Self identified as formal or informal family caregivers
* Over 18 years old
* Chinese
* Cantonese speaking

Exclusion Criteria:

* Cognitive disability
* Domestic helpers or maids
* Non Chinese

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2011-06; Primary Completion 2012-08 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Distress level | Change of distress level at pre-discharged(base-line) and 2 weeks and 4 weeks and 8 weeks post intervention
  Effect of telephone intervention on distress level measured at pre-discharged(baseline) and 2 weeks and 4 weeks and 8 weeks post intervention .

SECONDARY OUTCOMES:
Burden of care | Measured at pre-discharged(base-line) and 2 weeks and 4 weeks and 8 weeks post intervention
  Effect of telephone intervention on burden of care measured at pre-discharged(baseline) and 2 weeks and 4 weeks and 8 weeks post intervention
Quality of life | Measured at pre-discharged(base-line) and 2 weeks and 4 weeks and 8 weeks post intervention
  Effect of telephone intervention at pre-discharged(base-line) and 2 weeks and 4 weeks and 8 weeks post intervention

CONTACTS AND LOCATIONS:
Overall Officials: N F Shum, Principal Investigator — Queen Mary Hospital, Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, China